CLINICAL TRIAL: NCT03490214
Title: Non-invasive Imaging of Muscle Structure in Duchenne Muscular Dystrophy as Diagnostic and Progression Marker Using Multispectral Optoacoustic Tomography
Brief Title: Non-invasive Imaging of Muscle Structure in Duchenne Muscular Dystrophy Using Multispectral Optoacoustic Tomography
Acronym: MSOT_DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 67_18 B
Record Dates: First submitted 2018-03-19; First posted 2018-04-06 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Duchenne Muscular Dystrophy; Muscular Dystrophies; Muscular Dystrophy, Duchenne
Keywords: Optoacoustics; MSOT; Multispectral Optoacoustic Tomography
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscular Dystrophia (Experimental): Multispectral Optoacoustic Tomography (MSOT) of muscles (left and right, total 8 sites) leg proximal: Musculus quadriceps, distal: Musculus triceps surae arm proximal: Musculus biceps, distal: Musculus brachioradialis
  Interventions: Device: Multispectral Optoacoustic Tomography
- Healthy Volunteer (Active Comparator): Multispectral Optoacoustic Tomography (MSOT) of muscles (left and right, total 8 sites) leg proximal: Musculus quadriceps, distal: Musculus triceps surae arm proximal: Musculus biceps, distal: Musculus brachioradialis
  Interventions: Device: Multispectral Optoacoustic Tomography

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography — Non-invasive transcutaneous imaging of subcellular muscle components

SUMMARY:
This pilot study aims to assess subcellular muscle structure in patients with Duchenne X-linked progressive Duchenne muscular dystrophy (DMD) in comparison to healthy volunteers using multispectral optoacoustic tomography (MSOT). During MSOT, a transducer is placed on the skin similar to a conventional sonography and instead of sound, energy is supplied to the tissue by means of light flashes. This leads to a constant change of minimal expansions and contractions (thermoelastic expansion) of individual tissue constituents or molecules. The resulting sound waves can then be detected by the same examination unit.

DETAILED DESCRIPTION:
Duchenne X-linked progressive Duchenne muscular dystrophy (DMD) is one of the most common progressive childhood muscle diseases with an incidence of 1 in 3500 male newborns and is associated primarily with decreased life expectancy. From the age of 4-5 years manifest motor problems in everyday life, typical signs of proximal muscle weakness, with lab-chemical increase of the muscle enzyme (creatinine kinase, CK). Within a few years, relevant muscle and tendon shortening leading to joint malpositions and instability, as well as scoliosis and loss of walking around the age of 10 are formed. Supportive therapies can not curatively affect complications and progression of the disease. Pathogenetically, there is a deficiency of dystrophin, a structural protein of the sarcolemma, which is caused by mutations (usually deletions) of the dystrophin gene (Xp21.3-p21.2). The result of dystrophin deficiency is a necrosis of muscle cells that are replaced by connective tissue and adipose tissue. Clinical scores (6-minute walk test, 6MWT) and MRI studies to characterize the degenerative changes of skeletal muscle in the early stages are available for the quantitative assessment of the disease progression as well as therapy effects, the significance of which is controversially discussed. However, the highly sensitive assessment of gene therapy effects (e.g., PTC 124) will become increasingly important in the future. Sensitive, non-invasive methods for the detection of early muscle degeneration and muscle function in the course are of great clinical and scientific importance. The purpose of this first pilot study is to investigate whether the differences in skeletal muscle composition of healthy volunteers and ambulatory patients with early stage DMD can be quantified and characterized using multispectral optoacoustic tomography (MSOT). This could in the future generate a completely new, non-invasive method to develop non-invasive biomarkers of disease progression or therapy response.

ELIGIBILITY:
DMD-Patients

Inclusion Criteria:

* Histologic or genetically proven DMD
* Age 3-10 years

Exclusion Criteria:

-

Healthy controls

Inclusion Criteria:

* Male
* Age 3-10 years

Exclusion Criteria:

* Suspected muscular disease/myopathia
* missing informed consent

Ages: 3 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Muscular lipid content | Single time point (1 day)
  Quantitative lipid signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD compared to healthy control Units: arbitrary units (a.u.)
Muscular collagen content | Single time point (1 day)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD compared to healthy control Units: arbitrary units (a.u.)

SECONDARY OUTCOMES:
Muscular myo-/hemoglobin content | Single time point (1 day)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD compared to healthy control Units: arbitrary units (a.u.)
Correlation of lipid signal with age/disease duration | Single time point (1 day)
  Quantitative lipid signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with individual disease duration/age (in month)
Correlation of myo-/hemoglobin signal with age/disease duration | Single time point (1 day)
  Quantitative moo-/hemoglobin signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with individual disease duration/age (in month)
Correlation of lipid signal with 6MWT | Single time point (1 day)
  Quantitative lipid signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with 6-minute walk test (6MWT, distance in meters, less distance means higher disease severity)
Correlation of lipid signal with MRC | Single time point (1 day)
  Quantitative lipid signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with Medical Research Council (MRC, scale: 0-5, lower score means less muscular strength, measured for each individual muscles) muscle scale
Correlation of collagen signal with 6MWT | Single time point (1 day)
  Quantitative collagen signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with 6-minute walk test (6MWT, distance in meters, less distance means higher disease severity)
Correlation of collagen signal with MRC | Single time point (1 day)
  Quantitative collagen signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with Medical Research Council (MRC, scale: 0-5, lower score means less muscular strength, measured for each individual muscles) muscle scale
Correlation of myo-/hemoglobin signal with 6MWT | Single time point (1 day)
  Quantitative myo-/hemoglobin signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with 6-minute walk test (6MWT, distance in meters, less distance means higher disease severity)
Correlation of myo-/hemoglobin signal with MRC | Single time point (1 day)
  Quantitative myo-/hemoglobin signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD correlated with Medical Research Council (MRC, scale: 0-5, lower score means less muscular strength, measured for each individual muscles) muscle scale
Signal differences left and right muscles | Single time point (1 day)
  Comparison of quantitative signal levels (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with DMD/healthy controls in right and left body muscular groups (upper and lower body)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, Dr., Principal Investigator — Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen; Regina Trollmann, Prof. Dr., Principal Investigator — Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen
Locations (1):
- Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Regensburger AP, Fonteyne LM, Jungert J, Wagner AL, Gerhalter T, Nagel AM, Heiss R, Flenkenthaler F, Qurashi M, Neurath MF, Klymiuk N, Kemter E, Frohlich T, Uder M, Woelfle J, Rascher W, Trollmann R, Wolf E, Waldner MJ, Knieling F. Detection of collagens by multispectral optoacoustic tomography as an imaging biomarker for Duchenne muscular dystrophy. Nat Med. 2019 Dec;25(12):1905-1915. doi: 10.1038/s41591-019-0669-y. Epub 2019 Dec 2. PMID 31792454